CLINICAL TRIAL: NCT05864677
Title: Efficacy of Cerebrolisin in the Prevention of Postoperative Delirium in Cardiac Surgery Patients
Brief Title: Cerebrolysin in Prevention of Postoperative Delirium in Cardiac Surgery
Acronym: Cereb-POD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Medical University of Lublin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KE-0254/235/11/2022
Record Dates: First submitted 2023-02-14; First posted 2023-05-18 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-05

CONDITIONS: Neurocognitive Disorders; Surgery-Complications; Critical Illness; Brain Damage; Cardiac Disease
MeSH Terms: conditions — Neurocognitive Disorders; Critical Illness; Brain Injuries; Heart Diseases | interventions — cerebrolysin

STUDY DESIGN:
Intervention Model Description: Adult patients undergoing CABG under general anesthesia will be included in this study. After signing informed consent patients will be randomized using a double-blinded envelope method into two groups: C - control and CER - patients receiving Cerebrolysin at the dose of 50 mL before surgery followed by 50 mL on the morning of days 1,2,3 and 4.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group S - standard treatment (No Intervention): Patients will be treated in accordance with the current recommendations. Patients with every postoperative complication (severe postoperative bleeding, wound infection, hemodynamically unstable) and those undergoing reoperation will be excluded from this study.
- Group CER - treatment with Cerebrolysin (Active Comparator): Patients will be treated in accordance with the current recommendations and receiving additional treatment with Cerebrolysin.
  Interventions: Drug: Cerebrolysin

INTERVENTIONS:
Drug: Cerebrolysin — Patients, who will be randomized to group CER, will receive Cerebrolysin at the dose of 50 mL before surgery, followed by 50 mL on the morning of days 1,2,3, and 4.
  Arms: Group CER - treatment with Cerebrolysin

SUMMARY:
Postoperative delirium (POD) and postoperative neuropsychological dysfunction are frequently noted in critically ill patients undergoing elective or emergency surgery and treated in the intensive care unit (ICU). Delirium is a serious complication that prolongs hospital stay and contributes to poor outcomes and increased risk of death. The pathomechanisms of delirium are still not very well recognized and there are several theories that seem to explain it. The most important pathomechanisms of delirium are associated with cerebral ischaemia, disorders in acetylcholinergic system, disorders in neuronal plasticity and oxidative stress. Cerebrolysin, a mixture of various peptides obtained from the structural proteins of the pig's brain, possesses strong antioxidative and neuronal protective properties. Cerebrolysin is recommended to treat patients with dementia, after cerebral ischemia and after brain trauma. It has been documented that Cerebrolysin reduces the severity of secondary brain damage after ischemia, improving neuronal plasticity and then cognitive function, and reducing severity of oxidative stress. Based on these properties it can be speculated that Cerebrolysin may reduce the risk of postoperative delirium in patients undergoing elective surgery, which are associated with a high risk of postoperative delirium.

DETAILED DESCRIPTION:
The main hypothesis: Cerebrolysin may be an effective drug to treat dementia and post-ischemic damage. It may improve neuronal plasticity, increase the activity of acetychocholinergic system, and reduces the severity of oxidative stress - all of them are the main factors corresponding to the risk of delirium.

The study will be conducted in accordance with the Declaration of Helsinki, after obtaining approval from the Bioethical Committee and signed informed consent from each patient eligible to participate in the study.

After signing informed consent patients will be randomized using a double-blinded envelope method into two groups: C - control and CER - patients receiving Cerebrolysin at the dose of 50 mL before surgery followed by 50 mL on the morning of days 1,2,3 and 4. The Montreal Cognitive Assessment (MoCA) scale and Mini-Mental State Examination Score (MMSE) will be performed a day before surgery to detect eventual neuropsychological disorders before surgery. The postoperative delirium will be detected with MoCA, MMSE and the Confusion Assessment Method for ICU (CAM-ICU) performed on day 5 after surgery. Additionally, 10 mL of plasma will be collected to assess the following neuro-biomarkers: S100β protein, neurofilament light protein (HNL), Tau protein, ubiquitin carboxy-terminal hydrolase L1 (UCH-L1), and myelin basic protein (MBP). All these biomarkers will be assessed pre-operatively (before Cerebrolysin administration) and on postoperative days 1, 3, and 5. Additionally, routine blood examinations such as arterial blood analysis, blood morphology with NLR and PLR, serum albumin, and CRP will be measured at the same time points.

ELIGIBILITY:
Inclusion Criteria:

* adult patients aged 18 - 90 years (male and female) undergoing elective coronary artery bypass graft surgery with cardiopulmonary bypass (extracorporeal circulation) not longer than 120 min.
* written informed consent,
* patients without a history of neurology diseases (stroke, cerebral trauma, treated for seizure),
* patients without stenosis of the carotid artery,

Exclusion Criteria:

* any neurological disease,
* intra-operative cardiac arrest,
* perioperative blood transfusion,
* cardiopulmonary bypass (extracorporeal circulation) longer than 120 min,
* any reoperation,
* lack of signed consent for this study,

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-01-15 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary end-point is to analyze changes in CAM-ICU test the incidence of delirium on the postoperative day 5. | baseline and 5 days
  The incidence of delirium will be primarily diagnosed with the CAM-ICU test. The CAM-ICU test will be performed one day before surgery (baseline) and on postoperative day 5. Delirium will be diagnosed if the patient's mental state changes from their baseline and/or fluctuation in mental status.
The primary end-point is to analyze changes in MoCA scale the incidence of delirium on the postoperative day 5. | baseline and 5 days
  The incidence of postoperative cognitive impairment will be diagnosed with the Montreal Cognitive Assessment Scale (MoCA) performed one day before surgery (baseline) and on postoperative day 5. Cognitive dysfunction will be diagnosed when patients score 22 or less on the MoCA scale. Patients who scored 22 or less before surgery will be excluded.
The primary end-point is to analyze changes in MMSE test the incidence of cognitive impairment on the postoperative day 5. | baseline and 5 days
  The incidence of postoperative cognitive impairment will be diagnosed with the Mini-Mental State Examination (MMSE) test performed one day before surgery (baseline) and on postoperative day 5. Cognitive dysfunction will be diagnosed when patients score 22 or less on the MMSE test. Patients who scored 22 or less before surgery will be excluded.

SECONDARY OUTCOMES:
The secondary end-points are the analysis of length of hospital stay. | one month after surgery.
  The length of hospital stay will be calculated in patients receiving Cerebrolysin and treated without Cerebrolysin. The length of hospital stay and outcome will be analyzed one month after surgery. All patients without postoperative delirium who required prolonged hospitalization (more than seven days) due to wound infection or cardiac arrhythmias will be excluded from this analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University, Lublin, Poland